CLINICAL TRIAL: NCT02084225
Title: Feasibility, Perceived Utility and Sustainability of Using Ultrasound-guided Regional Anesthesia by Local Providers in a Limited Resource Conflict Setting
Brief Title: Ultrasound Guided Regional Anesthesia for Acute Injury in Low Resource Settings
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Salmon, Margaret, M.D. (Individual)
Collaborators: Sonosite/Fuji Film - (in kind) (Unknown); The ultrasound for the study was given to the sites by Sonosite/Fuji but the company (Unknown); had no other role in the study. (Unknown); MedShare - (in kind) (Unknown); The needles and syringes and kit contents were given to the sites by MedShare but the (Unknown); company had no role in the study. (Unknown)
Responsible Party: Principal Investigator, margaret salmon, Global Health Emergency Medicine, University Health Network, Toronto General Hospital, Salmon, Margaret, M.D.
Other Study IDs: NB0001
Record Dates: First submitted 2014-03-09; First posted 2014-03-11 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Pain Management; Acute Injuries
Keywords: low resource; conflict setting; ultrasound guided regional anesthesia; acute injuries; pain management; education; ultrasound; trauma; emergency department
MeSH Terms: conditions — Agnosia; Wounds and Injuries; Emergencies | interventions — Lidocaine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Course participants: Physicians, nurses and orthopedic officers who staff the emergency intake and orthopedic procedure area of HEAL hospital, Goma DRC, Black Lion Hospital, Addis Ababa and Kindu General Hospital in Kindu DRC. These participants recorded their nerve block intervention over one year for pain management and assessed patient pain level after 10 cc lidocaine.
  Interventions: Procedure: ultrasound guided regional nerve block

INTERVENTIONS:
Procedure: ultrasound guided regional nerve block — participants were the physicians performing the procedure
  Other Names: lidocaine 1% and 2%

SUMMARY:
The purpose of this study is to determine feasibility, perceived utility and sustainability of training local providers in ultrasound guided regional anesthesia for acute pain management in a limited-resource conflict setting.

DETAILED DESCRIPTION:
To the investigators knowledge, this is the first study of feasibility, perceived utility and sustainability of USRA as a pain management tool in a low-resource conflict setting and is one of the only large studies to date to assess USRA by local providers for emergent pain relief due to injury in patients presenting to an acute care center.

ELIGIBILITY:
Inclusion Criteria:

* participants were chosen by hospital administration

Exclusion Criteria:

* only chosen participants were included

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants include medical doctors and orthopedic or trauma nurses (officers) who staff the emergency department and/or orthopedic procedure area where acute injuries are treated.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Participant perceived utility of ultrasound guided nerve block | study start - ongoing (24 months)
  Participants filled out a data sheet on each block performed. The participant stated yes/no if a block was found to have positive utility

SECONDARY OUTCOMES:
Participant course satisfaction | at course end (5 days)
  Post course evaluation of course satisfaction and balance of didactic simulation and clinical scanning

OTHER OUTCOMES:
Patient pain reduction (VAS) | up to 18 months
  Pain reduction was calculated using 1 - 10 of a VAS. The patients was asked to rate pain before and 20 minutes after the procedure
Post procedure serious and non serious adverse event | before and up to 48 hours after every block performed
  Patients were followed up to 48 hours post procedure in order to monitor for adverse events including residual nerve sensory deficit and/or infection at the injection site
Indication for use of USRA by participant | up to 18 months of study period
  Participants recorded patient indication for offering USRA when presenting with acute injury including burns gun shot wounds lacerations, bone injuries soft tissue injuries and painful dressing changes

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Salmon, MD MPH, Principal Investigator — HEAL Hospital
Locations (3):
- Black Lion Hospital, Addis Ababa, Ethiopia
- Republic of the Congo (2):
  - HEAL Hospital, Goma
  - John Maurice Kikuni Salmu, Kindu